CLINICAL TRIAL: NCT00464009
Title: Development and Evaluation of a Medical Intervention for Early Childhood Caries
Acronym: IMB-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: R. Gary Rozier, DDS, UNC-CH School of Public Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-P-91251/4-02
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2009-09

CONDITIONS: Early Childhood Dental Caries
Keywords: Early childhood caries - ECC; Prevention; Continuing medical education; Randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Group A practices (n=39) received didactic training and course materials in oral health screening, referral, counseling and application of fluoride varnish.
  Interventions: Behavioral: Continuing medical education
- B (Active Comparator): Group B practices (n=41) received the same as Group A and were offered weekly conference calls providing advice and support.
  Interventions: Behavioral: Continuing medical education
- C (Active Comparator): Group C practices (n=41) received the same as Group B and were also offered in-office follow-up visits providing hands-on advice and support.
  Interventions: Behavioral: Continuing medical education

INTERVENTIONS:
Behavioral: Continuing medical education — Group A practices took part in a 90 minute lecture with slides, case-based presentations and discussions of the clinical interventions, instruction in children's dental development, common dental diseases and prevention, screening, referral, counseling and fluoride varnish application. Group B practices received the same as group A and additionally were offered support through telephone conference calls using "learning collaborative" methods where staff receive ongoing support from CME instructors and learn from one another as they begin to implement systems for preventive care in their practices. The conference calls were moderated by research staff with clinical expertise in primary health care who had assisted in other interventions among NC pediatric and family medicine offices. Group C received the same intervention as Group B and were offered additional in-office support for implementation of preventive dental procedures provided by a dental hygienist.

SUMMARY:
This study aimed to evaluate the effect of three forms of continuing medical education (CME) on provision of preventive dental services to Medicaid-enrolled children by medical personnel in primary care physician offices.

DETAILED DESCRIPTION:
Practice-based, randomized controlled trial. Setting: 1,400 pediatric and family physician practices in North Carolina providing care to an estimated 240,000 Medicaid-eligible children aged 0-3 years. Interventions: Group A practices (n=39) received didactic training and course materials in oral health screening, referral, counseling and application of fluoride varnish. Group B practices (n=41) received the same as Group A and were offered weekly conference calls providing advice and support. Group C practices (n=41) received the same as Group B and were offered in-office visit providing hands-on advice and support. Outcome measures were computed from reimbursement claims submitted to NC Division of Medical Assistance. Primary outcome measure: rate of preventive dental services provision per 100 well-child visits. Secondary outcome measure: % of practices providing 20 or more preventive dental visits.

ELIGIBILITY:
Inclusion Criteria:

* pediatric or family physician Medicaid practice in North Carolina

Exclusion Criteria:

* participation in related pilot study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-02; Primary Completion 2002-04 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Rate of preventive dental services provision per 100 well-child visits. | One year following initial training.

SECONDARY OUTCOMES:
Percent of practices providing 20 or more preventive dental visits. | One year following initial training.

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Rozier, DDS, Principal Investigator — UNC-CH, School of Public Health, Department of Health Policy and Administration
Locations (1):
- UNC-CH, School of Public Health, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Quinonez RB, Pahel BT, Rozier RG, Stearns SC. Follow-up preventive dental visits for Medicaid-enrolled children in the medical office. J Public Health Dent. 2008 Summer;68(3):131-8. doi: 10.1111/j.1752-7325.2007.00055.x. PMID 18179471
- [Result] Rozier RG, Sutton BK, Bawden JW, Haupt K, Slade GD, King RS. Prevention of early childhood caries in North Carolina medical practices: implications for research and practice. J Dent Educ. 2003 Aug;67(8):876-85. PMID 12959161
- [Result] Slade GD, Rozier RG, Zeldin LP, Margolis PA. Training pediatric health care providers in prevention of dental decay: results from a randomized controlled trial. BMC Health Serv Res. 2007 Nov 2;7:176. doi: 10.1186/1472-6963-7-176. PMID 17980021
- [Result] Rozier RG, Slade GD, Zeldin LP, Wang H. Parents' satisfaction with preventive dental care for young children provided by nondental primary care providers. Pediatr Dent. 2005 Jul-Aug;27(4):313-22. PMID 16317972